CLINICAL TRIAL: NCT00067691
Title: Acupuncture for Shortness of Breath in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001029-01 (NIH)
Record Dates: First submitted 2003-08-25; First posted 2003-08-27 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Lung Neoplasms; Breast Neoplasms
Keywords: Lung cancer; Breast cancer; Shortness of breath; Dyspnea; Metastasis; Breathlessness; Acupuncture
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Dyspnea; Neoplasm Metastasis | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The purpose of this study is to determine whether acupuncture is effective in relieving shortness of breath among breast and lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of local or metastatic breast or lung cancer
* Shortness of breath with onset after cancer diagnosis
* Life expectancy of at least 4 weeks

Exclusion Criteria:

* Prior acupuncture
* Other conditions suspected of causing shortness of breath, such as congestive heart failure, sarcoid disease, pneumonia, or obesity
* No chest wall deformity
* Neuromuscular disorders
* Pulmonary vascular disease
* Anemia
* Uncontrolled pain or infection
* Heart valve dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-11; Study Completion 2003-11

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan-Kettering Institute for Cancer Research, New York, New York, United States